CLINICAL TRIAL: NCT04459702
Title: A Phase IIa Randomized, Controlled Study of Combination Therapies to Treat COVID-19 Infection
Brief Title: A Study of Combination Therapies to Treat COVID-19 Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Was never started
Sponsor: ProgenaBiome (Other)
Collaborators: Big Corona Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-043
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: COVID; COVID-19; Corona Virus Infection; Coronavirus Infection; Coronavirus Sars-Associated as Cause of Disease Classified Elsewhere; Coronavirus-19; SARS-CoV 2; SARS Pneumonia
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine; Azithromycin; Ritonavir; Lopinavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual Therapy (Experimental): Dual Therapy utilizing hydroxychloroquine and azithromycin.
  Interventions: Drug: hydroxychloroquine; Drug: Azithromycin
- Quadruple Therapy (Experimental): Quadruple therapy utilizing hydroxychloroquine, lopinavir, ritonavir, and azithromycin
  Interventions: Drug: hydroxychloroquine; Drug: Azithromycin; Drug: Ritonavir; Drug: Lopinavir

INTERVENTIONS:
Drug: hydroxychloroquine — Treatment with the drug hydroxychloroquine
  Other Names: Plaquenil
Drug: Azithromycin — Treatment with the drug azithromycin
  Other Names: Zithromax
Drug: Ritonavir — Treatment with the drug ritonavir
  Other Names: norvir
  Arms: Quadruple Therapy
Drug: Lopinavir — Treatment with the drug lopinavir
  Arms: Quadruple Therapy

SUMMARY:
This study seeks to determine whether dual or quadruple therapy is more effective in treating COVID-19.

DETAILED DESCRIPTION:
In this study, patients will be administered either dual or quadruple therapy and have PCR tests run daily to determine efficacy as indicated by time to non-infectivity

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the subject understands the procedures required for the study and the purpose of the study
2. Healthy, ambulant male or female subjects 18 years of age to 65 years of age
3. Positive test for COVID-19 by RT-PCR at screening
4. Subjects must agree to practice at least one highly effective method of birth control for the duration of the study. This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. Subjects not of reproductive potential will be exempt (e.g. post-menopausal, surgically sterilized)
5. Subjects must agree they will do their best to attend the treatment facility daily for 10 days

Exclusion Criteria:

1. Refusal to sign informed consent form
2. Negative test for COVID-19 by RT-PCR at screening
3. Severe disease symptomatically including pneumonia, respiratory distress, tachypnea, shortness of breath, temperature > 38 degrees; pleuritic pain, or frequent cough.
4. Known drug allergy to any of the investigational medications
5. Currently taking medication with known drug interactions with investigational medications (listed in appendix)
6. Prescription or other antiviral medications
7. Any comorbidities which constitute health risk for the subject
8. Pregnant or lactating females;
9. weight < 110lb;
10. porphyria
11. established retinal disease
12. Inability to attend daily for 10 days
13. Any contraindications for treatment with hydroxychloroquine

    1. Hypoglycemia
    2. Known G6PD deficiency
    3. Porphyria
    4. Anemia
    5. Neutropenia
    6. Alcoholism
    7. Myasthenia gravis
    8. Skeletal muscle disorders
    9. Maculopathy
    10. Changes in visual field
    11. Liver disease
    12. Psoriasis
    13. History of QT >500msec
    14. History of torsades de pointes
14. Anemia from pyruvate kinase and G6PD deficiencies
15. Abnormal EKG with QT prolongation acquired or from birth
16. History of jaundice or high fevers prior to developing COVID-19
17. Treatment with any of the medications listed in Appendix II
18. Treatment with any anti-epileptic medication
19. Treatment with any other drug not listed that affects the QT interval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Treatment by Reduced Symptoms NEWS (National Early Warning System) scores | 6 months
  Time to reduced symptoms in each treatment group as indicated by NEWS scores, which rate patient status based on a zero to three scale for 8 parameters. These values are added up to create the NEWS score. The lower the NEWS score, the better the patient's clinical condition. Zero is the lowest possible score, whereas 7 or greater represents a high degree of clinical risk.
Efficacy of Treatment by Time to Non-Infectivity | 10 days
  Time to non-infectivity as measured by PCR testing

SECONDARY OUTCOMES:
Safety of Dual Therapy as Measured by Symptoms rated on the NEWS (National Early Warning System) sores | 6 months
  Patient symptoms will be recorded using the NEWS system, which rates patient status based on a zero to three scale for 8 parameters. These values are added up to create the NEWS score. The lower the NEWS score, the better the patient's clinical condition. Zero is the lowest possible score, whereas 7 or greater represents a high degree of clinical risk.
Safety of Quadruple Therapy as Measured by Symptoms rated on the NEWS (National Early Warning System) scores. | 6 months
  Patient symptoms will be recorded using the NEWS system, which rates patient status based on a zero to three scale for 8 parameters. These values are added up to create the NEWS score. The lower the NEWS score, the better the patient's clinical condition. Zero is the lowest possible score, whereas 7 or greater represents a high degree of clinical risk.
Safety of Dual Therapy as Measured by Complete Blood Count | 6 months
  Changes in blood parameters measured in a Complete Blood Count (CBC).
Safety of Quadruple Therapy as Measured by Complete Blood Count | 6 months
  Changes in blood parameters measured in a Complete Metabolic Panel.
Safety of Dual Therapy as Measured by Metabolic Panel -Albumin | 6 months
  Changes in serum albumin levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Albumin | 6 months
  Changes in serum albumin levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - A/G Ratio | 6 months
  Changes in serum albumin/globulin ratio
Safety of Dual Therapy as Measured by Metabolic Panel A/G Ratio | 6 months
  Changes in serum albumin/globulin ratio
Safety of Quadruple Therapy as Measured by Metabolic Panel - Alkaline Phosphatase | 6 months
  Changes in serum alkaline phosphatase levels
Safety of Dual Therapy as Measured by Metabolic Panel Alkaline Phosphatase | 6 months
  Changes in serum alkaline phosphatase levels
Safety of Dual Therapy as Measured by Metabolic Panel - AST | 6 months
  Changes in serum AST levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - AST | 6 months
  Changes in serum AST levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - ALT | 6 months
  Changes in serum ALT levels
Safety of Dual Therapy as Measured by Metabolic Panel ALT | 6 months
  Changes in serum ALT levels
Safety of Dual Therapy as Measured by Metabolic Panel BUN/Creatinine Ratio | 6 months
  Changes in serum BUN/Creatinine Ratio
Safety of Quadruple Therapy as Measured by Metabolic Panel BUN/Creatinine Ratio | 6 months
  Changes in serum BUN/Creatinine Ratio
Safety of Quadruple Therapy as Measured by Metabolic Panel - BUN | 6 months
  Changes in serum Blood Urea Nitrogen levels
Safety of Dual Therapy as Measured by Metabolic Panel - BUN | 6 months
  Changes in serum Blood Urea Nitrogen levels
Safety of Dual Therapy as Measured by Metabolic Panel - Calcium | 6 months
  Changes in serum calcium levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Calcium | 6 months
  Changes in serum calcium levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Carbon Dioxide | 6 months
  Changes in serum carbon dioxide levels
Safety of Dual Therapy as Measured by Metabolic Panel - Carbon Dioxide | 6 months
  Changes in serum carbon dioxide levels
Safety of Dual Therapy as Measured by Metabolic Panel - Chloride | 6 months
  Changes in serum chloride levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Chloride | 6 months
  Changes in serum chloride levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Creatinine | 6 months
  Changes in serum creatinine levels
Safety of Dual Therapy as Measured by Metabolic Panel - Creatinine | 6 months
  Changes in serum creatinine levels
Safety of Dual Therapy as Measured by Metabolic Panel - Globulin | 6 months
  Changes in serum globulin levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Globulin | 6 months
  Changes in serum globulin levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Glucose | 6 months
  Changes in blood glucose levels
Safety of Dual Therapy as Measured by Metabolic Panel - Glucose | 6 months
  Changes in blood glucose levels
Safety of Dual Therapy as Measured by Metabolic Panel - Potassium | 6 months
  Changes in blood potassium levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Potassium | 6 months
  Changes in blood potassium levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Total Bilirubin | 6 months
  Changes in serum total bilirubin levels
Safety of Dual Therapy as Measured by Metabolic Panel - Total Bilirubin | 6 months
  Changes in serum total bilirubin levels
Safety of Dual Therapy as Measured by Metabolic Panel - Total Protein | 6 months
  Changes in serum total protein levels
Safety of Quadruple Therapy as Measured by Metabolic Panel - Total Protein | 6 months
  Changes in serum total protein levels
Safety of Dual Therapy as Measured by Treatment Related SAE | 6 months
  Presence or absence of treatment related serious adverse events Grade III or higher
Safety of Quadruple Therapy as Measured by Treatment Related SAE | 6 months
  Presence or absence of treatment related serious adverse events Grade III or higher

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome; Thomas Borody, MD, PhD,, Principal Investigator — Big Corona Ltd.
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No